CLINICAL TRIAL: NCT05806203
Title: Randomized Controlled Trial for Use of Low Intensity Shockwave for Patients With Dyspareunia
Brief Title: A Study of Participants Ages 21-65 Diagnosed With Dyspareunia and the Effects of Low Intensity Shockwave Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SoftWave Tissue Regeneration Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018453-1
Record Dates: First submitted 2023-02-21; First posted 2023-04-10 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Female Dyspareunia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Low Intensity plus PT (Active Comparator): Participants receive active low intensity shockwave treatment from plus typical physical therapy.
  Interventions: Device: Low intensity shockwave treatment to pelvic floor region plus typical physical therapy
- Sham Shockwave Treatment plus PT (Sham Comparator): Participant receives sham shockwave treatment plus typical physical therapy.
  Interventions: Device: Sham shockwave treatment plus typical physical therapy

INTERVENTIONS:
Device: Low intensity shockwave treatment to pelvic floor region plus typical physical therapy — Treatment dose: 1,000 - 1,500 shocks, 2.5-3.0 Hz, 0.06-0.10 mJ/mm2 (Intensity of 6-8), 8 to 12 minutes
  Arms: Low Intensity plus PT
Device: Sham shockwave treatment plus typical physical therapy — Inactive dose of shockwave treatment
  Arms: Sham Shockwave Treatment plus PT

SUMMARY:
Dyspareunia is defined as a complaint of persistent or recurring pain or discomfort associated with attempted or complete vaginal penetration

e purpose of this study is to determine the effectiveness of low intensity shockwave treatment for patients with dyspareunia and their ability to tolerate sexual activity, (i.e., penetration of vagina, self or partnered pleasure).

Participants will:

* Be given a preliminary physical therapy examination and evaluation.
* Be asked to attend weekly low intensity shockwave treatment visits.
* Be asked to complete 3 Month follow up questionnaires

DETAILED DESCRIPTION:
This study seeks to determine the effectiveness of low intensity shockwave (LiSWT) for patients with dyspareunia, with the primary objective being the ability to tolerate penetration of the vagina and sexual activity, (self or partnered pleasure). A secondary objective of the study is an improved quality of life.

This is a single blind, randomized controlled trial, with randomized placebo phase design.

A total of 60 participants enrolled at 4 clinical sites will be blinded to the group they are assigned to, (treatment or sham). Clinical investigators cannot be blinded to treatment or sham in order to deliver the treatment.

There are two arms of the study: the Intervention arm where subjects receive active low intensity shockwave treatment plus typical physical therapy. Intervention is the delivery of shockwaves to the pelvic floor region using Softwave Tissue RegenerationTechnologies OrthoGold 100 MTS OP155 unfocused parabolic probe electrohydraulic device.

The Control arm subjects receive sham shockwave treatment plus typical physical therapy.

Each clinical site will have an envelope with pre-determined even and odd numbers determining randomization. Upon enrollment a random number from the envelope will be drawn and assigned to the participant.

At 4-6 weeks participants in the control arm will be given the option of moving to the shockwave (intervention) arm. Participants will spend 4 to 4 1/2 months in the study receiving treatment once per week, 4-6 weeks duration for both treatment arms. Subjects will then be contacted for a 3-month follow-up by phone completing their study participation.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of dyspareunia (pain with intercourse and/or vaginal penetration)
* Cisgender female or have natal vaginal tissu
* Has not started hormonal therapy within the past 2 weeks
* Has not received pelvic floor physical therapy within the past 2 weeks
* Is able to electronically access informed consent and outcomes measures forms

Exclusion Criteria:

* Have a diagnosis of lichen sclerosis
* Have an active infection (e.g. herpes)
* Are earlier than 12 weeks post-surgery
* Are earlier than 6 weeks postpartum
* Have a history of gynecological cancer
* Have a history of pelvic radiation
* Are actively undergoing cancer treatments
* Are currently pregnant
* Currently using lidocaine or cortisone

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender female or have natal vaginal tissue
Enrollment: 60 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Tampon Test | up to 6 weeks
  A self-reported measurement of pain on a numeric scale from 0 to 10, with 0 signifying no pain and 10 signifying extreme pain.
Numerical pain rating scale for tampon test | up to 6 weeks
  A self-reported measurement of pain on a numeric scale from 1 to 10, with 0 signifying no pain and 10 signifying extreme pain.
Female Sexual Function Index, (FSFI) | up to 6 weeks
  A validated, self-reported questionnaire assessing different domains of female sexual function including desire, arousal, lubrication, orgasm, satisfaction, and pain. Scores range from 2.0 to 36.0. Lower scores indicate greater risk of female sexual dysfunction, and higher scores indicate better outcomes in overall sexual function.

SECONDARY OUTCOMES:
Numeric pain score for deep penetration. | Completed once per week for 4 to 6 weeks
  A self-reported measurement of pain on a numeric scale from 1 to 10, with 0 signifying no pain and 10 signifying extreme pain.
Beck Depression Scale | Completed once per week for 4 to 6 weeks
  Sel-reported scale consisting of 21 items of emotional, behavioral, and somatic symptoms. Scoring ranges from 0, (no symptoms) to 27, (severe symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Roberts, Principal Investigator
Locations (1):
- New You Health and Wellness, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No